CLINICAL TRIAL: NCT01959854
Title: Evaluation of Xanthan Gum Eye Drops in Patients With Dry Eye
Brief Title: Efficacy of Topical 0.2% Xanthan Gum in Patients With Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SIFI SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XNTME2013
Record Dates: First submitted 2013-10-07; First posted 2013-10-10 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- carboxymethylcellulose (Active Comparator): 1 drop in each eye four times a day for 30 days
  Interventions: Device: carboxymethylcellulose
- xanthan gum (Experimental): 1 drop in each eye four times a day for 30 days
  Interventions: Device: xanthan gum

INTERVENTIONS:
Device: carboxymethylcellulose — 0.25% carboxymethylcellulose preservative free
  Other Names: THERADROP
  Arms: carboxymethylcellulose
Device: xanthan gum — 0.2% xanthan gum preservative free
  Other Names: OXISTOP
  Arms: xanthan gum

SUMMARY:
The purpose of this study is to evaluate the effect of an ophthalmic solution containing 0.2% xanthan gum in reducing symptoms and signs of dry eye as well as tear film markers of oxidative stress.

DETAILED DESCRIPTION:
Oxidative stress is the result of an imbalance between the production of reactive oxygen species (ROS) and antioxidant systems . The eye is constantly exposed to solar UV radiation which is the major inducer of ROS production and therefore oxidative stress has been implicated in the pathogenesis of several eye disease, including dry eye. Xanthan gum is a complex exopolysaccharide utilized as a food additive. Its chemical structure shows a capacity to react with ROS indicating a role as an anti-oxidative molecule.

In the present study aging patients with dry eye will be enrolled. Signs and symptoms of dry eye as well as levels of oxidative stress in tear will be evaluated afte 30 days of treatment with eye drops containing carboxymethylcellulose or xanthan gum.

ELIGIBILITY:
Inclusion Criteria:

* Ocular Surface Disease Index > 12<23 and age >59 yrs

Exclusion Criteria:

* contact lens wear and use of other ophthalmic solutions with the exception of artificial tears

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Ocular surface disease index (OSDI) | change from baseline OSDI at 30 days
  OSDI is a questionnaire including 12 questions to be asked to the patient. From the questionnaire it will be possible to calculate the OSDI score which is a reliable and valid measurement for dry eye severity.

SECONDARY OUTCOMES:
Visual analogue rating scale (VARS) | change from baseline VARS at 30 days
  Global symptoms of dry eye will be graded by patients using a 0-100 mm visual analogue rating scale (0 = no symptoms to 100 = severe symptoms)
Fluorescein staining | change from baseline staining at 30 days
  Eye surface damage (corneal and conjunctival) assessed by fluorescein staining will be graded against standard chart (Oxford system)

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Aragona, MD, Principal Investigator — University of Messina (ITALY)
Locations (1):
- University of Messina, Messina, Italy